CLINICAL TRIAL: NCT00526513
Title: Study of Safety and Effectiveness of Apidra® in Combination With Basal Insulin in Patients With Type 1 & 2 Diabetes Mellitus
Acronym: SCALE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APIDR_L_01913
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Insulin Glulisine — subcutaneous injection of insulin glulisine at meal, 1 to 3 injections a day based on the condition of the patient in addition to a basal SC insulin injection at bedtime

SUMMARY:
Primary Objectives:

To determine the effect of insulin glulisine on glycemic control (HbA1c, FBG & PPBG) from baseline to the end of the study.

Secondary Objectives:

To evaluate the safety of insulin glulisine in basal/bolus regimen by monitoring the incidence of hypoglycemia and other adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or type 2 diabetes mellitus previously treated for 6 months with prandial insulin + Basal insulin or Premix (Type I) or by either a basal insulin + OAD or basal + RHI/other short acting analogue insulin or Premix (Type II) with HbA1c >7%.
* Adequate hepatic and renal functions
* Ability and willingness of a tight antidiabetic therapy and to perform blood glucose self-monitoring and especially blood glucose profiles, using a blood glucometer at home.

Exclusion Criteria:

* Pregnant or lactating women or women of childbearing potential not using adequate contraception.
* Patients with hypersensitivity to insulin glulisine or to any of the excipients.
* History of diabetic ketoacidosis.
* Diabetic retinopathy with surgical treatment (laser photocoagulation or vitrectomy) in the 3 months prior to study entry or which may require surgical treatment within 3 months of study entry.
* Alcohol abuse or drug abuse.
* Clinically relevant cardiovascular, gastrointestinal, hepatic, neurological, endocrine, hematological or psychiatric illness, other serious illnesses, uncontrolled medical conditions or active infections making implementation of the protocol difficult.
* Medical, psychiatric, or neurologic condition that renders the patient unable to understand the nature and scope of the study. Mental retardation or language barrier such that the patient is unable to give informed consent.
* Participation in an investigational trial within 30 days of study entry.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Glycosylated Haemoglobin (HbA1c) | At 3 months after the treatment start
Glycosylated Haemoglobin (HbA1c) | At 6 months after the treatment start

SECONDARY OUTCOMES:
Control of Fasting Blood Glucose (FBG) | At 3 months after the treatment start
Control of Post-Prandial Glycemia (PPBG) | At 3 months after the treatment start
Control of Post-Prandial Glycemia (PPBG) | At 6 months after the treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Mosaad I Morsi, MBBCH, MSC, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Cairo, Egypt